CLINICAL TRIAL: NCT07249606
Title: Real-world Observation of Momelotinib Effectiveness in Myelofibrosis (ROME)
Brief Title: Momelotinib Effectiveness in Myelofibrosis
Status: Not yet recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: MPN0325
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Myelofibrosis (MF)
Keywords: Myelofibrosis; momelotinib; real-world; post polycythemia; post essential thrombocythemia
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MF patients treated with momelotinib: Patients diagnosed with primary or post-polycythemia vera/post-essential thrombocythemia myelofibrosis treated with momelotinib according to clinical practice from AIFA authorization.

SUMMARY:
Observational study aimed at evaluating the use of momelotinib in patients with primary or post polycythemia vera (PV) or post essential thrombocythemia myelofibrosis (post-ET MF) in a real-world setting.

DETAILED DESCRIPTION:
This is a multicenter prospective and retrospective observational clinical study in adult patients with primary or post polycythemia vera (PV) or post essential thrombocythemia myelofibrosis (post-ET MF) being treated with momelotinib in a real-world setting. The aim of the study is to evaluate the efficacy of momelotinib in terms of splenic response. All patients are managed according to the clinical practice of the participating Center.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older.
2. Patients diagnosed with primary or post-polycythemia vera/post-essential thrombocythemia myelofibrosis start treatment with MMB according to clinical practice from AIFA authorization.
3. Patients with palpable splenomegaly at baseline of momelotinib treatment.
4. Informed consent signed, if applicable.

Exclusion Criteria:

1. Diagnosis of MPN, unclassifiable, myelodysplastic/myeloproliferative neoplasms, myelodysplastic syndromes, essential thrombocythemia, polycythemia vera.
2. Accelerated/blast phase of MF.
3. Patients with platelets <20 x10(9)/L at baseline of MMB treatment.
4. Patients JAK inhibitors-exposed for other diseases apart from MF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for primary myelofibrosis or post polycythemia vera or post essential thrombocythemia at the Italian hemathology units with access to momelotinib. All participating centers belong to the GIMEMA network.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2028-01-02 (Estimated); Study Completion 2028-04-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy of momelotinib in splenic response improving | Six months
  To assess the splenic response in terms of rate of patients with more or equal than 50% palpatory reduction compared to baseline at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Passamonti, Principal Investigator — Ematologia, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milano

IPD SHARING:
Plan to Share IPD: No